CLINICAL TRIAL: NCT02752347
Title: An Electromyography Study Comparing the Impact of Using RMEs on Muscle Activity Among Growing Orthodontic Patients (A Prospective Clinical Study)
Brief Title: An Electromyography Study Comparing the Impact of Using RMEs on Muscle Activity Among Growing Orthodontic Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riyadh Colleges of Dentistry and Pharmacy (Other)
Responsible Party: Principal Investigator, Nancy Ajwa, Resident, Riyadh Colleges of Dentistry and Pharmacy
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: FPGRP/43534001/14
Record Dates: First submitted 2016-04-15; First posted 2016-04-27 (Estimated); Last update posted 2017-10-09 (Actual); Status verified 2017-10

CONDITIONS: Malocclusion
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- unilateral crossbite (Experimental): unilateral crossbite patients with constricted maxilla, going to be treated by rapid maxillary expanders the surface Electromyography (surface EMG device) device will be used to examine the muscle activities before and after expansion
  Interventions: Device: Surface EMG device
- control (No Intervention): the surface Electromyography (surface EMG device) device will be used to examine the muscle activities on normal patients
- Bilateral crossbite (Experimental): Bilateral crossbite patients with constricted maxilla, going to be treated by rapid maxillary expanders the surface Electromyography (surface EMG device) device will be used to examine the muscle activities before and after expansion
  Interventions: Device: Surface EMG device

INTERVENTIONS:
Device: Surface EMG device — measuring the muscles activity using surface EMG device
  Other Names: BioRadio EMG Device
  Arms: Bilateral crossbite; unilateral crossbite

SUMMARY:
Compare the impact of using rapid maxillary expanders on masticatory muscle activities (Masseter and Anterior Temporalis muscles) among different posterior cross-bite patient (unilateral, bilateral) as well as compare the cross-bite side and non-cross-bite sides of the same preadolescent unilateral crossbite patient before the expansion and after one month of the completion treatment period using surface electromyography device.

DETAILED DESCRIPTION:
Compare the impact of using rapid maxillary expanders on masticatory muscle activities (Masseter and Anterior Temporalis muscles) between the cross-bite side and non-cross-bite sides of the same preadolescent orthodontic patient before the expansion and after one month of the completion treatment period.

Two channels surface Electromyography sEMG (BioRadio), will be position to record the activity of anterior temporal (AT) and masseter (MM) muscles in three different statuses:

* Rest → patients will instruct to not bite on his/her teeth.
* Clench → patients will instruct to made a maximum voluntary clench on cotton rolls positioned around the first molar, for 5 sec "the cotton clench", and a maximum voluntary clench without the interposed rolls for 5 sec "the "clench".

  * This procedure followed the Sforza et al. protocol.
* During function "mastication" → The patients will instruct to chew on a chewing gum for 20 sec (20 continuous masticatory cycles).

Examination frequency:

The patients will be examined two times as follow:

Test 1: Immediately before rapid maxillary expanders cementation, Test 2: 5 months later (1 month after the retention phase).

the same procedure will be done on 35 patients (control group)

ELIGIBILITY:
Inclusion Criteria:

1. Uni-lateral/ or bilateral posterior cross-bite.
2. Patients with erupted permanent maxillary and mandibular first molars.
3. Will be treated by rapid maxillary expanders, (the appliance planning to be worn for approximately 5 months).
4. Age ranged from 9 to 12.
5. Males and females.
6. Not under any medications.
7. Skeletal Class I or Class II (based on ANB angle, convexity, and Wits appraisal).
8. No active caries.
9. Healthy periodontal tissues.
10. Subjects with no signs of TMD or condylar problems.

Exclusion Criteria:

1. History of any functional appliance treatment.
2. Oral, systemic disease or any syndromes.
3. Patients under any medications.

6. Patients with symptoms of Temporomandibular disorders. 4. Neuropathic conditions. 5. Open and deep-bite.

Ages: 9 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-06 (Actual); Study Completion 2017-12-30 (Estimated)

PRIMARY OUTCOMES:
measuring the masticatory muscles activity using electromyography device | Test 1: before cementation of rapid maxillary expander, Test 2: after removal of rapid maxillary expander by 1 month
  the muscle activities of masticatory muscles using surface Electromyography device before and compare it after the maxillary expansion using Rapid Maxillary Expanders (to study the impact of the expanders on the muscles), the muscle activity will be in form of micro volt/second (mV/sec), the data will aggregated then exported on excel sheet in a form of numbers for statistical analysis

CONTACTS AND LOCATIONS:
Overall Officials: Hezekiah A Mosadomi, DMD, Study Chair — Riyadh Colleges of Dentistry and Pharmacy
Locations (1):
- Riyadh Colleges of Dentistry and Pharmacy, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
data will be used for a research purpose only , will not be shared with any other institution